CLINICAL TRIAL: NCT05252208
Title: Is Stretching Superior to Aerobic Training for Reducing Blood Pressure?
Brief Title: Stretching vs Walking for Lowering Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2874
Record Dates: First submitted 2022-02-12; First posted 2022-02-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Parallel groups: Two groups: Walking exercise and stretching exercise
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching (Experimental): Stretching
  Interventions: Other: Stretching exercise
- Walking (Experimental): Walking
  Interventions: Other: Walking exercise

INTERVENTIONS:
Other: Stretching exercise — Stretching (30-45 minutes, 5 days per week, 6 months)
  Arms: Stretching
Other: Walking exercise — Walking (30-45 minutes, 5 days per week, 6 months)
  Arms: Walking

SUMMARY:
High blood pressure is a leading risk factor for cardiovascular disease. Traditionally, one of the ways to treat or prevent high blood pressure is to prescribe aerobic exercise training (i.e. brisk walking). Stretching may also be effective because it may cause changes in blood vessel stiffness and therefore reduce resistance to blood flow. The study will assess a group of individuals (i.e. 96) participating in a supervised stretching or walking program five days per week for six months to determine whether stretching is superior for reducing blood pressure. This research will contribute to recommendations about the most effective exercise programs for reducing blood pressure and risk of cardiovascular disease.

DETAILED DESCRIPTION:
Hypertension or high blood pressure is a prevalent and leading risk factor for heart disease and stroke afflicting seven million people in Canada and costing our health system approximately $20 billion annually. The prevailing exercise recommendation for people with hypertension is to perform aerobic training (i.e. brisk walking) as a non-pharmacological way to moderately reduce blood pressure. Evidence from several recent studies indicates flexibility training may accrue more positive changes in blood pressure than aerobic training. Additional recent studies show stretching can reduce arterial stiffness and sympathetic nervous system activation, suggesting physiological mechanisms by which blood pressure might be reduced through exercises designed mostly to improve flexibility. The purpose of this study is to determine if a 6-month flexibility program is superior to aerobic training for reducing 24-hour blood pressure measurements, improving measures of vascular function (i.e. arterial stiffness), and improving the ratio of parasympathetic to sympathetic nervous system activation. This study involves a randomized controlled trial of 96 men and women presenting with either high-normal blood pressure (systolic 130 to 139 mmHg or diastolic 85 to 89 mmHg) or stage 1 hypertension (systolic 140 to 159 mmHg or diastolic 90 to 99 mmHg) stratified by blood pressure (i.e. either high normal or stage 1 hypertension), sex, and age (≥55y or <55y) and randomized to one of two groups for six months duration: 1) a flexibility program (30 minutes of stretching per day); or 2) an aerobic training program (30 minutes of brisk walking per day). Assessments pre- and post-intervention and three months later include: 24-hour ambulatory blood pressure, arterial stiffness, and heart rate variability. .

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure between 130 and 159 mmHg OR diastolic blood pressure between 85 and 99 mmHg
* Able to walk unaided for 30 minutes
* Can safely perform exercises as determined by the Get Active Questionnaire

Exclusion Criteria:

* Not on blood pressure medication unless it has been a stable dose for 6 months and target blood pressure has not been achieved (i.e. below 140/90 mmHg)
* Smoking
* Already performing 150 minutes or more moderate to vigorous physical activity per week
* Already involved in a flexibility-training program (e.g. Yoga or Pilates)
* Pregnant or lactating or planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Night time systolic and diastolic blood pressure | Change from baseline night time blood pressure at 6 months
  Blood pressure assessed during the night with an automated device

SECONDARY OUTCOMES:
Day time systolic and diastolic blood pressure | Change from baseline day time blood pressure at 6 months
  Blood pressure assessed during the day with an automated device
Sitting systolic and diastolic blood pressure | Change from baseline sitting blood pressure at 6 months
  Blood pressure assessed while sitting
Lying systolic and diastolic blood pressure | Change from baseline lying blood pressure at 6 months
  Blood pressure assessed while lying supine
Arterial stiffness | Change from baseline arterial stiffness at 6 months
  Arterial stiffness assessed with aplanation tonometry
Heart rate variability | Change from baseline heart rate variability at 6 months
  Heart rate variability assessed with electrocardiography
Hamstrings flexibility | Change from baseline hamstrings flexibiliity at 6 months
  Hamstrings flexibility assessed with a sit-and-reach test
Shoulder flexibility | Change from baseline shoulder flexibility at 6 months
  Shoulder flexibility assessed with a goniometer
Peak oxygen consumption | Change from baseline peak oxygen consumption at 6 months
  Peak oxygen consumption assessed with a metabolic cart during a progressive-intensity treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No